CLINICAL TRIAL: NCT05742087
Title: Study of the Consequences of Anti-GFAP Antibodies on the Peripheral Nervous System
Brief Title: Neuropathy and Anti-GFAP Antibodies
Acronym: Neuro-GFAP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5018
Record Dates: First submitted 2022-12-01; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Neurological Diseases or Conditions; Neurological Diseases Associated to Anti GFAP Antibodies
Keywords: GFAP; neuropathy
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting with neurological symptoms and anti-GFAP antibodies in the CSF.: This is a non-interventional study involving biological samples. Samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "iological Resource Center of the Hospices Civils de Lyon" (CRB-HCL) (including tissue, cells or biological fluids).
  The group will be composed of patients included in the French cohort of patients with neurological syndromes and anti-GFAP antibodies in the CSF.
  Interventions: Other: Clinical examination; Other: electroneuromyography (ENMG)

INTERVENTIONS:
Other: Clinical examination — The examination performed by the clinician of the patient will be analyzed from the cohort as previously explained.
Other: electroneuromyography (ENMG) — Data from the ENMGs will be extracted from the cohort and analyzed.

SUMMARY:
Anti-Glial Fibrillary Acidic Protein (GFAP) are antibodies associated to inflammatory diseases of the central nervous system. The GFAP protein is highly expressed by astrocytes explaining these syndromes, but GFAP is also expressed by immature and non-myelinating Schwann cells. Thus, these antibodies could also lead to damages of the peripheral nervous system (PNS). Moreover, such damages have already been reported on small studies, and there is a need for larger cohorts.

The investigators will use the cohort of patients with neurological syndromes and anti-GFAP antibodies identified in the cerebrospinal fluid (CSF) of the "Reference center for paraneoplastic neurological syndromes and autoimmune encephalitis" to determine the frequency of the PNS involvement in these patients.

ELIGIBILITY:
Inclusion Criteria:

* - Age > 18 years old
* Neurological symptoms
* Anti-GFAP antibodies identified in the CSF

Exclusion Criteria:

* - Uncomplete data in the medical records of patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 patients presenting with neurological symptoms and with identified anti-GFAP antibodies in the CSF, included in the French cohort of patients with neurological syndroms and anti-GFAP antibodies identified in the cerebrospinal fluid (CSF) of the "Centre de reference des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes", will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Cranial nerves abnormality at clinical examination of abnormal ENMG | Immediately after diagnosis
  Data concerning the clinical examination and the ENMG will be extracted from the cohort of patients with neurological syndroms and anti-GFAP antibodies identified in the cerebrospinal fluid (CSF) of the "Centre de reference des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes".

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites autoimmunes, Lyon, France